CLINICAL TRIAL: NCT03645356
Title: Evaluation of the Efficacy of Clear Aligners in the Correction of Severe Dental Crowding Cases Combined With Premolar Extraction Versus Vestibular Fixed Orthodontic Appliances: A Randomized Clinical Controlled Trial
Brief Title: Comparison Between Clear Aligners and Traditional Fixed Appliances in the Treatment of Four-premolar-extraction Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-07-2018
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Malocclusion, Angle Class I; Malocclusion; Displaced or Missing Teeth; Crowding
MeSH Terms: conditions — Malocclusion, Angle Class I; Malocclusion; Anodontia; Crowding | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fixed appliances (Active Comparator): patients will be treated using fixed appliances in order to align their teeth after extraction of four premolars
  Interventions: Device: Fixed Appliances
- clear aligners (Experimental): patients will be treated using clear aligners in order to align their teeth after extraction of four premolars
  Interventions: Device: Clear Aligners

INTERVENTIONS:
Device: Fixed Appliances — Using an MBT-prescription of metallic brackets, patients will be treated in the conventional way
  Arms: fixed appliances
Device: Clear Aligners — Using a sequence of clear aligners, patients will be give an aligner every two weeks until the completion of treatment
  Arms: clear aligners

SUMMARY:
Patients who have severe crowding that require four premolars extraction will be treated in this study. The efficacy of the clear aligners and vestibular fixed appliances will be assessed. The treatment result of these two different methods will be explored using the Peer Assessment Rating (PAR) in two different times (T0: Before treatment, T1: After treatment) and the American Board of Orthodontics Objective Grading System (ABO-OGS) after treatment (T1).

There are two groups:

First group (Experimental): the patients in this group will be treated using clear aligners.

Second group (Control): the patients in this group will be treated using fixed appliances.

DETAILED DESCRIPTION:
For years, orthodontists and dentists have used removable appliances for orthodontic treatment. Today, with the CAD/CAM technology, clear aligners treat a broader range of cases with greater precision. They consist of a series of plastic aligners that are intended to replace conventional wire and bracket technology for many orthodontic cases. Each custom manufactured aligner exerts gentle, continuous forces to move teeth incrementally from their original state to a final, treated state. Each aligner is worn for about two weeks, then replaced by the next in the series until the final position is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Class I malocclusion with severe crowding (more than 5 mm of tooth-size-arch-length-discrepancy).
* Good oral hygiene and periodontal health.
* No severe skeletal discrepancy.
* Normal proclination for the upper and lower incisors.
* No congenitally missing or extracted teeth (except for the third molars).
* No history of previous trauma to the maxillofacial region or surgical interventions.

Exclusion Criteria:

* Bimaxillary dentoalveolar severe protrusion.
* Previous orthodontic treatment.
* Subject with psychological abnormalities.
* Subject with systemic diseases.
* Subject has known allergy to latex and plastic

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-19 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change in the American Board of Orthodontics - Objective Grading System (ABO-OGS) | T1: one day before the commencement of treatment. T2: one day following the end of treatment (that is expected to happen within 24 months)
  Eight domains are evaluated:
  Alignment: No more than 2 points shall be subtracted for any tooth when it is poorly aligned; Marginal Ridges: The total number of deductions shall be subtracted from 32 to give the score for this domain; Buccolingual inclination: If the mandibular lingual cusps or maxillary buccal cusps are more than 1 mm from the straight edge surface, 1 point shall be subtracted for that tooth; Occlusal Contacts: If a cusp is out of contact with the opposing arch, 1 point is subtracted for that tooth; Occlusal relationships. The total number of deductions are subtracted from 24 to give the score for occlusal relationships; Overjet; Interproximal contacts. If no interproximal spaces exist, then no points are subtracted; and Root angulation: Any deviations in roots' angulations will cause a deduction form the general score. Finally, a case that loses more than 30 points will be considered a failure. A case that loses less than 20 points will be considered acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Samer T Jaber, DDS MSc, Principal Investigator — PhD Student in Orthodontics, University of Damascus Dental School, Damascus; Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bollen AM, Huang G, King G, Hujoel P, Ma T. Activation time and material stiffness of sequential removable orthodontic appliances. Part 1: Ability to complete treatment. Am J Orthod Dentofacial Orthop. 2003 Nov;124(5):496-501. doi: 10.1016/s0889-5406(03)00576-6. PMID 14614415
- [Background] Drake CT, McGorray SP, Dolce C, Nair M, Wheeler TT. Orthodontic tooth movement with clear aligners. ISRN Dent. 2012;2012:657973. doi: 10.5402/2012/657973. Epub 2012 Aug 14. PMID 22928114
- [Background] Giancotti A, Di Girolamo R. Treatment of severe maxillary crowding using Invisalign and fixed appliances. J Clin Orthod. 2009 Sep;43(9):583-9; quiz 582. No abstract available. PMID 19904051
- [Background] Hennessy J, Al-Awadhi EA. Clear aligners generations and orthodontic tooth movement. J Orthod. 2016 Mar;43(1):68-76. doi: 10.1179/1465313315Y.0000000004. PMID 25939782
- [Background] Kravitz ND, Kusnoto B, BeGole E, Obrez A, Agran B. How well does Invisalign work? A prospective clinical study evaluating the efficacy of tooth movement with Invisalign. Am J Orthod Dentofacial Orthop. 2009 Jan;135(1):27-35. doi: 10.1016/j.ajodo.2007.05.018. PMID 19121497
- [Background] Li W, Wang S, Zhang Y. The effectiveness of the Invisalign appliance in extraction cases using the the ABO model grading system: a multicenter randomized controlled trial. Int J Clin Exp Med. 2015 May 15;8(5):8276-82. eCollection 2015. PMID 26221410
- [Background] Zhang XJ, He L, Guo HM, Tian J, Bai YX, Li S. Integrated three-dimensional digital assessment of accuracy of anterior tooth movement using clear aligners. Korean J Orthod. 2015 Nov;45(6):275-81. doi: 10.4041/kjod.2015.45.6.275. Epub 2015 Nov 20. PMID 26629473